CLINICAL TRIAL: NCT00125515
Title: Evaluation of NMDA Antagonist for Opiate Dependence
Brief Title: Memantine and Naltrexone Treatment for Opioid Dependence
Acronym: NAMHS-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #4847/R01-15822; K23DA000429 (NIH)
Record Dates: First submitted 2005-07-28; First posted 2005-08-01 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Opioid Dependence
Keywords: Heroin; Opiates; naltrexone; memantine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Memantine; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo plus oral naltrexone
  Interventions: Drug: Naltrexone
- Memantine 30 mg bid (Active Comparator): Memantine 30 mg bid plus oral naltrexone
  Interventions: Drug: Memantine; Drug: Naltrexone
- Memantine 15 mg bid (Active Comparator): memantine 15 mg bid plus oral naltrexone
  Interventions: Drug: Memantine; Drug: Naltrexone

INTERVENTIONS:
Drug: Memantine — One arm receives 30 mg bid and the other arm receives receives 15mg bid
  Arms: Memantine 15 mg bid; Memantine 30 mg bid
Drug: Naltrexone — Patients received the equivalent of 50 mg/day. Dispensed as 100 mg on Mondays and Wednesdays and 150 mg on Fridays.

SUMMARY:
The goal of this study is to test the efficacy of memantine (a noncompetitive NMDA receptor antagonist) as an adjunct to the maintenance treatment with naltrexone in detoxified heroin-dependent individuals.

DETAILED DESCRIPTION:
The primary aim of this study is to test the efficacy of memantine, a noncompetitive NMDA receptor antagonist, in reducing early attrition and improving outcome in opioid-dependent individuals maintained on naltrexone.

This double-blind, 12-week trial will include heroin-dependent patients who completed detoxification. Participants will be randomly assigned to one of three conditions: naltrexone and placebo, naltrexone and memantine (15 mg bid), or naltrexone and memantine (30 mg bid). Naltrexone will be taken 3 times each week at the clinic, while memantine or placebo will be taken at home. In addition, twice each week patients will receive a psychosocial intervention that will include motivational interviewing and cognitive-behavioral relapse prevention. The goal of the psychosocial intervention is to improve compliance with medication and maintain abstinence. Baseline assessments will be taken and compared to those completed at study visits, which will occur 3 times each week.

ELIGIBILITY:
Inclusion:

* Adult, aged 18-60.
* Meets DSM-IV criteria for current opiate dependence disorder of at least six months duration, supported by a positive urine for opiates and a positive naloxone challenge test if the diagnosis is unclear.
* Able to give informed consent.

Exclusion:

* Pregnancy or breastfeeding
* Failure in a sexually active woman to use adequate contraceptive methods
* Active medical illness that might make participation hazardous, such as untreated hypertension, acute hepatitis with SGOT or SGPT levels > 2 times normal, unstable diabetes, or chronic organic mental disorder (e.g., AIDS dementia)
* Active psychiatric disorder that might interfere with participation or make participation hazardous, including DSM-IV schizophrenia, bipolar disorder with mania or psychosis, and depressive disorder with suicide risk or 1 or more suicide attempts within the past year.
* History of allergic reaction to buprenorphine, naloxone, memantine, naltrexone, clonidine, or clonazepam
* Currently prescribed or regularly taking opiates for chronic pain or medical illness
* Current participation in another intensive psychotherapy or substance abuse treatment program or currently prescribed psychotropic medications
* Current participation in a methadone maintenance treatment program and/or regular use of illicit methadone ( > 30 mg per week)
* History of accidental drug overdose in the last 3 years or any other significant history of overdose following detoxification, defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2005-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, M.D., Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: stars website — http://stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals who applied for treatment at the Columbia University's Substance Treatment and Research Service outpatient clinic in New York City were recruited for this study.
Pre-assignment Details: Following consent participants were admitted to an inpatient unti at NYSPI for the purpose od detoxification and naltrexone induction. On the second day of induction they were randomized to a study arm.
Period: Overall Study
Arm/Group | Placebo | Memantine 30 mg Bid | Memantine 15 mg Bid
Started | 27 | 27 | 27
Completed | 7 | 7 | 6
Not Completed | 20 | 20 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Memantine 30 mg Bid | Memantine 15 mg Bid | Total
Number analyzed (Participants) | 27 | 27 | 27 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 27 | 81
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (9.6) | 42.0 (10.3) | 41.5 (9.4) | 41.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 3 | 15
  Male | 20 | 22 | 24 | 66
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 27 | 81

OUTCOME MEASURES:

1. Primary Outcome: Retention in Treatment
Description: The number of participants who were retained and completed all 12 weeks of treatment and study participation were compared between the three study groups.
Time Frame: Number of participants who complete 12 weeks of treatment
Population: All analysis were conducted based on intent-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Placebo | Memantine 30 mg Bid | Memantine 15 mg Bid
Number analyzed (Participants) | 27 | 27 | 27
participants | 7 | 5 | 6
Statistical Analysis 1: Comparison: Placebo vs Memantine 30 mg Bid vs Memantine 15 mg Bid; all statistical analysis were two tailed and employed an alpha significance level of 0.05; Test type: Superiority or Other; p = 0.32, Chi-squared

ADVERSE EVENTS:
Arm/Group | Placebo | Memantine 30 mg Bid | Memantine 15 mg Bid
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 1/27
Other Adverse Events (participants affected / at risk) | 16/27 | 17/27 | 10/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Memantine 30 mg Bid (N=27) | Memantine 15 mg Bid (N=27)
heroin overdose (General disorders) | 0 (0) | 0 (0) | 1 (1) — Overdose requiring hospitalization following relapse to heroin use.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Memantine 30 mg Bid (N=27) | Memantine 15 mg Bid (N=27)
headache (General disorders) | 5 (5) | 3 (3) | 2 (2)
insomnia (General disorders) | 7 (7) | 9 (9) | 8 (8)
body aches (General disorders) | 2 (2) | 2 (2) | 1 (1)
dizziness (General disorders) | 3 (3) | 2 (2) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1)
weakness (General disorders) | 1 (1) | 1 (1) | 3 (3)
diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 2 (2)
GI distress (Gastrointestinal disorders) | 7 (7) | 7 (7) | 0 (0)

LIMITATIONS AND CAVEATS:
It is possible that concomitant naltrexone might have exacerbated protracted withdrawal, thus masking the potential ameliorative effects of memantine that have been previously observed in other trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No